CLINICAL TRIAL: NCT06431776
Title: An Open-label, Multicenter Clinical Study to Evaluate the Efficacy and Safety of Inhaled Molgramostim in Pediatric Participants With Autoimmune Pulmonary Alveolar Proteinosis (aPAP).
Brief Title: Inhaled Molgramostim in Pediatric Participants With Autoimmune Pulmonary Alveolar Proteinosis (aPAP).
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Savara Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAV006-04
Record Dates: First submitted 2024-05-22; First posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Autoimmune Pulmonary Alveolar Proteinosis
Keywords: alveolar proteinosis; autoimmune; lung lavage; GM-CSF; children
MeSH Terms: conditions — Pulmonary Alveolar Proteinosis, Acquired; Pulmonary Alveolar Proteinosis | interventions — molgramostim; Colony-Stimulating Factors; regramostim

STUDY DESIGN:
Intervention Model Description: Open-label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- molgramostim (Experimental): Molgramostim 300 mcg administered once daily via nebulizer for 48 weeks.
  Interventions: Drug: Molgramostim

INTERVENTIONS:
Drug: Molgramostim — Molgramostim nebulizer solution will be administered once daily using a proprietary nebulizer optimized for the delivery of high molecular weight biologic compounds.
  Other Names: Recombinant human granulocyte-macrophage colony stimulating factor (rhGM-CSF).

SUMMARY:
The goal of this open-label study is to study molgramostim as a treatment for autoimmune pulmonary alveolar proteinosis (aPAP) in pediatric patients between age 6 and 18. The main questions it aims to answer are:

The effect of molgramostim on breathing tests and activity in pediatric patients with aPAP and the safety of molgramostim in pediatric patients with aPAP.

This is an open-label study: all participants will receive treatment with molgramostim.

Patients will:

* Take molgramostim once daily via nebulizer every day for 12 months.
* Visit the clinic approximately every 12 weeks for checkups and tests.
* Keep a diary of any oxygen use.

DETAILED DESCRIPTION:
This is an interventional open-label, single arm, multi-center study in pediatric subjects, age 6 through 18 years, who are diagnosed with autoimmune pulmonary alveolar proteinosis (aPAP).

The diagnosis of aPAP should be confirmed by an anti-GM-CSF antibody test and a history compatible with PAP based on patient symptoms, high resolution computed tomography of the lung, lung biopsy or bronchoalveolar lavage cytology.

The study consists of a 4-week screening period followed by a 48-week open-label treatment period. After completing the 48-week treatment or early withdrawal, subjects will enter a 4-week safety follow up period. The maximum treatment duration is 48-weeks, and the maximum study period will be 56 weeks. During the trial, lung lavage will be allowed as a rescue treatment in case of worsening of aPAP.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥6 and <18 years of age, at the time of signing the informed consent and informed assent (if applicable).
* Have a history of pulmonary alveolar proteinosis, based on examination of a lung biopsy, bronchoalveolar lavage cytology, or a high-resolution computed tomogram of the chest.
* Have a positive serum anti-GM-CSF autoantibody test result confirming aPAP.
* Have a hemoglobin (Hb)-adjusted diffusing capacity of the lung for carbon monoxide (DLCO) ≤70% predicted at Screening.

Exclusion Criteria:

* Have a diagnosis of hereditary (congenital) or secondary PAP, or a metabolic disorder of surfactant production.
* Have undergone treatment with Lung Lavage (WLL) within 1 month of Baseline

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
DLCO | 24 weeks
  Change in Hb-adjusted % predicted DLCO from Baseline.

SECONDARY OUTCOMES:
DLCO | 48-weeks
  Change in Hb-adjusted % predicted DLCO from Baseline .
6-minute walk distance | 24-weeks
  Absolute change from Baseline in 6-minute walk distance (6MWD)
6-minute walk distance | 48-weeks
  Absolute change from Baseline in 6-minute walk distance (6MWD).
PedsQL | 24-weeks
  Change from Baseline in Pediatric Quality of Life (PedsQLTM) Generic Core Scale score.
PedsQL | 48-weeks
  Change from Baseline in Pediatric Quality of Life (PedsQLTM) Generic Core Scale score.
Oxygen Saturation (SpO2) | 24 weeks
  Absolute change from Baseline in oxygen saturation (SpO2)
Oxygen Saturation (SpO2) | 48 weeks
  Absolute change from Baseline in oxygen saturation (SpO2)

OTHER OUTCOMES:
Adverse Events | 48 weeks
  Adverse events (AEs), including clinically significant findings on pulmonary function tests and safety laboratory assessments and adverse events of special interest (AESIs; hypersensitivity and chest pain).
Anti-GM-CSF Ab titer | 0, 4, 12,24,48 and 52 weeks
  Titers of anti-GM-CSF antibodies
FEV1 | 24 and 48-weeks
  Change from Baseline in forced expiratory volume in one second (FEV1) (% predicted)
FVC | 24 and 48-weeks
  Change from Baseline in Forced vital capacity (FVC) (% predicted)

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine Wasfi, MD, Ph.D., Study Director — Savara Inc.
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No